CLINICAL TRIAL: NCT01788566
Title: A Single-Arm, Multicenter, Open-Label, Phase 2 Study of Gemcitabine-Cisplatin Chemotherapy Plus Necitumumab (IMC-11F8) in the First-Line Treatment of Patients With Stage IV Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Gemcitabine-Cisplatin Chemotherapy Plus Necitumumab in the First-Line Treatment of Participants With Squamous Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14789; I4X-MC-JFCK (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — necitumumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Cisplatin + Necitumumab (Experimental): Necitumumab administered intravenously (IV) 800 milligram (mg) on Days 1 and 8 of each 3-week cycle.
  Gemcitabine administered IV at 1250 milligram per square meter (mg/m^2) on Days 1 and 8 of each 3 week cycle for a maximum of 6 cycles.
  Cisplatin administered IV at 75 mg/m^2 on Day 1 of each 3 week cycle for a maximum of 6 cycles.
  Interventions: Drug: Necitumumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Necitumumab — Administered IV
  Other Names: IMC-11F8; LY3012211; Portrazza®
Drug: Gemcitabine — Administered IV
  Other Names: Gemzar®; LY188011
Drug: Cisplatin — Administered IV

SUMMARY:
The purpose of this study is to see how participants with late stage lung cancer do on gemcitabine-cisplatin chemotherapy plus necitumumab. The study will also see how safe the drugs are in combination and to see how long the medicine stays in the body. The study will last approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous Non-small Cell Lung Cancer (NSCLC)
* Stage IV disease at time of study entry based on American Joint Committee on Cancer 7th edition
* Measurable disease at time of study entry as defined by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1
* Required to have a performance status (PS) 0-1

Exclusion Criteria:

* Nonsquamous NSCLC
* Prior anticancer therapy with monoclonal antibodies, signal transduction inhibitors, or any therapies targeting the epidermal growth factor receptor (EGFR), vascular endothelial growth factor (VEGF), or VEGF receptor
* Previous chemotherapy for NSCLC
* Major surgery or received any investigational therapy in the 4 weeks prior to study enrollment
* Chest irradiation within 12 weeks prior to randomization (except palliative irradiation of bone lesions, which is allowed)
* Brain metastases that are symptomatic or require ongoing treatment with steroids or anticonvulsants (participants who have undergone previous radiotherapy for brain metastases, who are now nonsymptomatic and no longer require treatment with steroids or anticonvulsants, are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deerfield Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Farmington Hills, Michigan
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris, France
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durango
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eindhoven
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Majadahonda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Started | 61
Completed | 53
Not Completed | 8
Not completed — Death | 4
Not completed — Adverse Event | 1
Not completed — Clinical Progressive Disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 49
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 48
  Asian | 11
  Black or African American | 1
  Missing | 1
Region of Enrollment [Number; unit: participants]
  Canada | 5
  Netherlands | 5
  United States | 11
  Taiwan | 8
  Mexico | 1
  France | 3
  Spain | 25
  Korea, Republic of | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) Objective Tumor Response Rate (ORR)
Description: ORR is confirmed best overall tumor response of CR or PR. According to RECIST v1.1, PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD; CR was defined as the disappearance of all target and non-target lesions. Percentage of participants was calculated as: total number of participants with a best tumor response of PR or CR among participants counted in the denominator/total number of participants treated with any amount of study drug, who has a complete radiographic assessment at baseline, and who has at least 1 complete radiographic assessment at postbaseline x 100%.
Time Frame: Baseline to Measured Progressive Disease (up to 17 Months)
Population: All participants who received any amount of study treatment and had evaluable baseline and postbaseline data for radiographic assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 54
Percentage of participants | 48.1 [34.34 to 62.16]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) duration is defined from the date of first dose of study drug to the date of death from any cause. OS was estimated by the Kaplan-Meier method. For participants who were not known to have died as of the data cut-off date, OS was censored at the date of last contact prior to the data cutoff date.
Time Frame: Baseline to Death from Any Cause (up to 17 Months)
Population: All participants who received any amount of study treatment. Participants censored=34.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 61
months | 11.7 [7.59 to NA] — The upper limit of the 95% confidence interval was not calculable due to the amount of censored data and immature survival data at the time of data cut-off.

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first dose of study drug until objective progressive disease (PD) or death for any cause. According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), PD was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the 20% relative increase, the sum must have also demonstrated an absolute increase of at least 5 millimeters (mm). The appearance of 1 or more new lesions was also considered progression. For participants not known to have died as of the data cut-off date and who do not have objective PD, PFS will be censored at the date of the last complete radiographic assessment.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause (up to 17 Months)
Population: All participants who received any quantity of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 61
months | 5.6 [3.68 to 6.87]

4. Secondary Outcome: Number of Participants Who Achieve Best Overall Disease Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD) [Disease Control Rate (DCR)]
Description: DCR is best overall response of SD, PR or CR. According to RECIST v1.1, PR defined as a ≥30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD; CR was defined as the disappearance of all target and non-target lesions. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started. Percentage of participants who achieved disease control = (those participants counted in the denominator with a best tumor response of SD, PR, or CR)/(the same denominator as for ORR)*100.
Time Frame: Baseline to Measured Progressive Disease or Participants Stops Study (up to 17 Months)
Population: All participants who received any quantity of study treatment and had evaluable baseline and postbaseline data for radiographic assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 54
percentage of participants | 81.5 [68.57 to 90.75]

5. Secondary Outcome: Percent Change in Tumor Size (CTS)
Description: CTS is defined as maximum percent improvement from baseline in the sum of target lesions.
Time Frame: Baseline until Measured Progressive Disease (up to 17 Months)
Population: All participants who received any quantity of study treatment and had evaluable baseline and postbaseline data for CTS.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 61
percent change | 39.68 (21.296)

6. Secondary Outcome: Pharmacokinetics (PK): Minimum (Cmin) Maximum Concentration (Cmax) of Necitumumab
Description: Pre-infusion Minimum Concentration (Cmin) and post-infusion (Cmax) necitumumab serum concentration
Time Frame: Predose Cycle 1 Day 8; Cycle 2 through 6 Day 1; End of Infusion (EOI) Cycle 1, 3, 5 Day 1
Population: All participants who received any amount of study treatment and had evaluable data for Cmax
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (ug/ml)
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 61
micrograms/milliliter (ug/ml)
  Predose Cycle 1 Day 8 | 70.8 (36.7)
  Predose Cycle 2 Day 1 | 67.5 (78.0)
  Predose Cycle 3 Day 1 | 106 (36.6)
  Predose Cycle 4 Day 1 | 115 (43.9)
  Predose Cycle 5 Day 1 | 141 (62.3)
  Predose Cycle 6 Day 1 | 126 (34.2)
  EOI Cycle 1 Day 1 | 266 (24.8)
  EOI Cycle 3 Day 1 | 352 (29.5)
  EOI Cycle 5 Day 1 | 360 (29.2)

7. Secondary Outcome: Number of Participants With Anti-Necitumumab Antibodies
Description: A participant was considered to have an anti-necitumumab antibody response if anti-drug antibodies (ADA) were detected at any time point. Treatment emergent antibodies were defined as any anti-necitumumab antibody titer equal to or greater than 4-fold the participant's baseline titer.
Time Frame: Baseline up to 30 Days Post Last Infusion (up to 17 Months)
Population: All participants who received any amount of study treatment and had evaluable baseline and postbaseline data for antibodies.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Number analyzed (Participants) | 61
participants
  Number of Participants with 1 Positive Titer | 9
  Treatment Emergent Antibody Positive | 4
  Neutralizing Antibody Detected | 3

ADVERSE EVENTS:
Arm/Group | Gemcitabine + Cisplatin + Necitumumab
Serious Adverse Events (participants affected / at risk) | 33/61
Other Adverse Events (participants affected / at risk) | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin + Necitumumab (N=61)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Malaise (General disorders) | 2 (3)
Pyrexia (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Catheter site abscess (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (2)
Diverticulitis (Infections and infestations) | 1 (2)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Conduct disorder (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Gemcitabine + Cisplatin + Necitumumab (N=61)
Anaemia (Blood and lymphatic system disorders) | 15 (38)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 19 (51)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (20)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Deafness (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Ototoxicity (Ear and labyrinth disorders) | 7 (14)
Tinnitus (Ear and labyrinth disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 3 (3)
Growth of eyelashes (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (10)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Cheilitis (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 20 (25)
Diarrhoea (Gastrointestinal disorders) | 18 (29)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 7 (7)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Lip dry (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 45 (79)
Odynophagia (Gastrointestinal disorders) | 2 (2)
Oesophageal pain (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 21 (44)
Vomiting (Gastrointestinal disorders) | 22 (39)
Asthenia (General disorders) | 25 (83)
Axillary pain (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Face oedema (General disorders) | 2 (2)
Fatigue (General disorders) | 22 (39)
Feeling cold (General disorders) | 2 (2)
Gait disturbance (General disorders) | 3 (3)
General physical health deterioration (General disorders) | 1 (1)
Influenza like illness (General disorders) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1)
Infusion site pain (General disorders) | 2 (2)
Infusion site urticaria (General disorders) | 1 (1)
Malaise (General disorders) | 5 (5)
Mucosal dryness (General disorders) | 2 (4)
Mucosal inflammation (General disorders) | 7 (9)
Non-cardiac chest pain (General disorders) | 4 (8)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 6 (7)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 12 (17)
Hypersensitivity (Immune system disorders) | 1 (1)
Adenoviral conjunctivitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (2)
Conjunctivitis (Infections and infestations) | 6 (11)
Dermatophytosis of nail (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Genital infection fungal (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (2)
Nail infection (Infections and infestations) | 2 (4)
Nasopharyngitis (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 12 (40)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1)
Scrotal infection (Infections and infestations) | 1/49 (1)
Skin infection (Infections and infestations) | 2 (3)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6)
Viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Blood urea increased (Investigations) | 1 (1)
Fibrin d dimer increased (Investigations) | 1 (1)
Glomerular filtration rate increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (11)
Platelet count decreased (Investigations) | 5 (11)
Platelet count increased (Investigations) | 3 (3)
Respiratory rate increased (Investigations) | 1 (1)
Troponin i increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 18 (24)
Weight increased (Investigations) | 5 (5)
White blood cell count decreased (Investigations) | 3 (3)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 35 (52)
Dehydration (Metabolism and nutrition disorders) | 5 (8)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 (45)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Aphasia (Nervous system disorders) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 14 (17)
Dysaesthesia (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 10 (12)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 4 (10)
Neurotoxicity (Nervous system disorders) | 4 (4)
Paraesthesia (Nervous system disorders) | 5 (8)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Confusional state (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 12 (14)
Irritability (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (2)
Micturition frequency decreased (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/49 (1)
Testicular pain (Reproductive system and breast disorders) | 1/49 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (24)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (14)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 12 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (25)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1)
Hair disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1/12 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1/49 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 28 (109)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 8 (15)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (11)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 3 (3)
Jugular vein distension (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days